CLINICAL TRIAL: NCT04897880
Title: A Phase II Study of Panobinostat in Pediatric, Adolescent and Young Adult Patients With Solid Tumors Including Osteosarcoma, Malignant Rhabdoid Tumor/Atypical Teratoid Rhabdoid Tumors and Neuroblastoma
Brief Title: A Study of Panobinostat in Pediatric Patients With Solid Tumors Including MRT/ATRT
Acronym: NORTH
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug supply
Sponsor: Australian & New Zealand Children's Haematology/Oncology Group (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); Secura Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACCT008/ASSG35; ACTRN12618000321246 (Registry Identifier: Australian New Zealand Clinical Trials Registry)
Record Dates: First submitted 2021-05-06; First posted 2021-05-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Rhabdoid Tumor; Atypical Teratoid/Rhabdoid Tumor; Malignant Rhabdoid Tumor; Recurrent Brain Tumor, Childhood
Keywords: Rhabdoid Tumor; Atypical Teratoid/Rhabdoid Tumor; Malignant Rhabdoid Tumor; Recurrent Brain Tumor, Childhood; Ashley; Pro00107447
MeSH Terms: conditions — Rhabdoid Tumor; Brain Neoplasms | interventions — Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Osteosarcoma [arm closed] (Experimental)
  Interventions: Drug: Panobinostat
- Malignant Rhabdoid Tumor/Atypical Teratoid Rhabdoid Tumor (Experimental)
  Interventions: Drug: Panobinostat
- Neuroblastoma [arm closed] (Experimental)
  Interventions: Drug: Panobinostat

INTERVENTIONS:
Drug: Panobinostat — Panobinostat capsules, 10mg, starting at a de-escalated dose of 8mg/m2 per day
  Other Names: Farydak®

SUMMARY:
This trial is evaluating the anti-tumor activity and side effects of panobinostat in treating patients with osteosarcoma, malignant rhabdoid tumor/atypical teratoid rhabdoid tumor (MRT/ATRT), and neuroblastoma.

DETAILED DESCRIPTION:
This is an open label, phase II, multi-centre study evaluating the anti-tumor activity of continuous, low dose of panobinostat in patients with recurrent or refractory solid tumors stratified by primary histology into osteosarcoma, malignant rhabdoid tumor/atypical teratoid rhabdoid tumor (MRT/ATRT), and neuroblastoma.

Patients will be stratified at study entry by tumor type into three strata: osteosarcoma, MRT/ATRT and neuroblastoma [osteosarcoma and neuroblastoma arms are closed to enrolment]. Patients will be enrolled onto the study following completion of their conventional therapy including chemotherapy and/or radiation treatment and completion of a three-week wash out period.

Panobinostat will then be administered as a continuous oral dose (starting at a de-escalated dose of 8mg/m2 per day), for up to 12 courses, a total of 48 weeks. The minimum dose is 2mg/m2 per day. Dosing will follow a dose de-escalation or escalation scheme for each stratum which will be determined by biological effect of the drug (measured in patient peripheral blood samples) and levels of toxicity (measured by dose limiting toxicity and adverse events observed). Dose levels for subsequent enrolments in each strata will be based on the de-escalated or escalated dose in each cohort. The final dose per strata will be that which achieves significant biological effect with acceptable toxicity that is maintained for a 4 week period.

Patients or their parents/guardians will be required to maintain a drug diary to monitor drug usage throughout the trial. Patients will be followed for up to 2 years from completion of study therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be < 40 years of age.
* Patient must have been histologically diagnosed with osteosarcoma, neuroblastoma or MRT/ATRT at time of diagnosis or relapse. [osteosarcoma and neuroblastoma arms are closed to recruitment].
* Patient disease is refractory to conventional therapy, in the case of osteosarcoma, neuroblastoma and MRT/ATRT or there is an absence of effective conventional therapy available in the case of ATRT. Patients must have stable disease (SD) or better following treatment with salvage therapy.
* Karnofsky performance level greater than or equal to 60% for patients 16 years of age and greater, OR Lansky performance levels greater than or equal to 60% for patients less than 16 years of age.
* Life expectancy of greater than 8 weeks.
* Fully recovered from acute toxic effects of all prior chemotherapy, immunotherapy or radiotherapy prior to entering study.
* Patients with CNS tumours who are receiving dexamethasone are on a stable/decreasing dose for at least 1 week.
* Adequate BM function
* Adequate renal function
* Adequate liver function
* Adequate cardiac function
* Adequate pulmonary function
* Adequate CNS function - seizure free for at least 2 months
* Adequate serum calcium, magnesium and potassium concentrations
* If female and post-menarchal, pregnancy test must be negative.
* If of reproductive potential, have agreed to use effective contraceptive method.
* If female and lactating, have agreed not to breastfeed.
* Patient and/or their legal guardian have signed a written informed consent form.

Exclusion Criteria:

* Have received myelosuppressive chemotherapy and/or biologic therapy within 3 weeks (4 weeks if prior nitrosourea).
* Have received local palliative radiotherapy within 2 weeks.
* Have received craniospinal radiotherapy within 3 weeks.
* Have received greater than or equal to 50% radiation of the pelvis within 6 weeks.
* Have received other substantial BM radiation within 6 weeks.
* Have received growth factor(s) within 1 week.
* Are receiving enzyme inducing anticonvulsant therapy.
* Are receiving medications associated with prolongation of QTc interval
* Are receiving hydrochlorothiazide.
* Are receiving metronidazole and/or disulfiram
* Have uncontrolled sepsis.
* Have previously received panobinostat.
* Have symptoms of congestive heart failure, uncontrolled cardiac rhythm disturbance, or a QTc greater than or equal to 450msec.

Max Age: 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
Event free survival | Up to 2 years after study enrolment
  Estimated 2-year Event free survival (EFS). EFS is calculated as the time from study enrolment to first documented disease progression, relapse or second malignancy, or death from any cause.
Overall Survival | Up to 2 years after study enrolment
  Estimated 2-year Overall Survival (OS). OS is calculated as the time from study enrolment to death from any cause.
Safety: Adverse events summarised by grade and type | From 1 week to 12 months after intervention commencement
  Graded and defined by CTCAE Version 4

SECONDARY OUTCOMES:
Efficacy as measured by Clinical Benefit Rate | At 6 and 12 months after intervention commencement
  Clinical benefit rate as the percentage of patients with stable disease or better using MRI/CT imaging).
  Stable disease is defined as MRT/ATRT/Osteosarcoma with CR/PR/MR/SD/ overall response.
  Neuroblastoma with CR/PR/SD or Non-CR/Non-PD overall response.

OTHER OUTCOMES:
Comparison between trial participants and historical control data | OS and EFS survival up to 2 years after study enrolment
  Comparing overall and event free survival for ATRT/MRT patients to historical data.

CONTACTS AND LOCATIONS:
Locations (11):
- The Preston Robert Tisch Brain Tumor Center, Duke University Medical Center, Durham, North Carolina, United States
- Australia (8):
  - John Hunter Children's Hospital, New Lambton, New South Wales
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Women's and Children's Hospital, North Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Monash Children's Hospital, Clayton, Victoria
  - The Royal Children's Hospital, Parkville, Victoria
  - Perth Children's Hospital, Nedlands, Western Australia
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-12-16): https://cdn.clinicaltrials.gov/large-docs/80/NCT04897880/SAP_000.pdf